CLINICAL TRIAL: NCT00551759
Title: A Phase II Study to Measure Response Rate and Toxicity of Neo-adjuvant Chemoradiotherapy With Oxaliplatin (OX) and Infusional 5-Fluorouracil (5-FU) Plus Cetuximab Followed by Post-Operative Docetaxel and Cetuximab in Patients With Operable Adenocarcinoma of the Esophagus
Brief Title: Chemotherapy, Radiation Therapy, and Cetuximab Followed by Surgery, Docetaxel, and Cetuximab in Treating Patients With Esophageal Cancer or Gastroesophageal Junction Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study used a two-stage design. After stage one, the study was terminated due to excess toxicity.
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000571857; U10CA021115 (NIH); E2205 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; chemoradiotherapy; oxaliplatin; cetuximab; docetaxel
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Fluorouracil; Oxaliplatin; Cetuximab; Docetaxel; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant therapy, Surgery, adjuvant therapy (Experimental): Neoadjuvant chemoradiotherapy and cetuximab: Patients (pts) receive oxaliplatin IV over 2 hours on days 1, 15, and 29, cetuximab IV over 1-2 hours on days 1, 8, 15, 22, and 29, and 5-FU IV over 24 hours on days 1-35. Pts also undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, and 29-33. Pts then proceed to surgery.
  Surgery: Pts undergo surgical resection within 4-8 weeks after completion of neoadjuvant chemoradiotherapy and cetuximab. Pts with an R0 or R1 resection proceed to adjuvant therapy. Pts whose tumors have not been completely resected or who have metastatic disease discontinue protocol therapy and receive further therapy at the discretion of the treating physician.
  Adjuvant therapy: Within 4-8 weeks after surgery, pts receive docetaxel IV over 1 hour on days 1, 8, 15, 22, and 29 and cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: Cetuximab; Drug: Docetaxel; Procedure: Surgery; Radiation: Radiotherapy

INTERVENTIONS:
Drug: 5-Fluorouracil — given IV
  Other Names: 5-FU; Fluorouracil; Adrucil; Efudex
Drug: Oxaliplatin — given IV
  Other Names: Trans-l-diaminocyclohexane oxalatoplatinum; Cis-[oxalato (trans-I-1,2-diaminocyclohexane) platinum(II)]; l-OHP; Eloxatin; Eloxatine; Dacplat; 5R96669
Drug: Cetuximab — given IV
  Other Names: Erbitux; C225
Drug: Docetaxel — given IV
  Other Names: Taxotere; RP 56976
Procedure: Surgery — Patients underwent surgical resection within 4-8 weeks after completion of neoadjuvant chemoradiotherapy and cetuximab.
Radiation: Radiotherapy — Patients underwent radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, and 29-33.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, fluorouracil, and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving these treatments before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving docetaxel and cetuximab after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving chemotherapy and radiation therapy together with cetuximab followed by surgery, docetaxel and cetuximab works in treating patients with esophageal cancer or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the pathologic complete response (pCR) rate of neoadjuvant chemoradiotherapy with OX/5-FU/radiotherapy (RT) plus cetuximab in patients with resectable adenocarcinoma of the esophagus.

Secondary

* To evaluate the safety of neoadjuvant chemoradiotherapy with OX/5-FU/RT plus cetuximab in patients with resectable adenocarcinoma of the esophagus.
* To evaluate the safety and tolerability of adjuvant therapy comprising cetuximab and docetaxel in these patients.
* To carry out exploratory studies to determine if activity of this regimen correlates with epidermal growth factor receptor (EGFR)-related genetic and pathway activation markers and circulating endothelial and tumor cells.

OUTLINE: This is a multicenter study.

* Neoadjuvant chemoradiotherapy and cetuximab: Patients receive oxaliplatin intravenously (IV) over 2 hours on days 1, 15, and 29, cetuximab IV over 1-2 hours on days 1, 8, 15, 22, and 29, and 5-FU IV continuously over 24 hours on days 1-35. Patients also undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, and 29-33. Patients then proceed to surgery.
* Surgery: Patients undergo surgical resection within 4-8 weeks after completion of neoadjuvant chemoradiotherapy and cetuximab. Patients with an R0 or R1 resection proceed to adjuvant therapy. Patients whose tumors have not been completely resected or who have metastatic disease discontinue protocol therapy and receive further therapy at the discretion of the treating physician.
* Adjuvant therapy: Within 4-8 weeks after surgery, patients receive docetaxel IV over 1 hour on days 1, 8, 15, 22, and 29 and cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, and then every 6 months for 3-5 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed adenocarcinoma of the esophagus (> 20 cm below the incisors) or gastroesophageal (GE) junction, untreated with chemotherapy, radiation therapy, and surgery. Endoscopy with biopsy and dilation was permitted.
* Tumor stage T2N0M0, T3N0M0, T1-3N+M0, or T1-3N0-1M1A as determined by imaging studies performed no greater than 4 weeks prior to registration, and biopsy, where appropriate. Celiac nodal metastasis (M1A disease) was permitted if other eligibility criteria were met. Data from endoscopic ultrasound and endoscopy were required for staging. The following imaging was required: CT scan with IV contrast and PET or PET+CT. If the PET/CT incorporates CT with IV contrast, then a separate CT is not required. If laparoscopy or other relevant procedures were performed, the data were to be incorporated into stage assignment. Any lesion suspicious for metastasis had to have been biopsied to prove eligibility.
* Tumor extension into cardia, if present, must have been no more than 2 cm.
* Tumors must have been considered surgically resectable (T1-3, not T4).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Granulocytes > 1,000/ mm³
* Platelets > 100,000 μL
* Creatinine normal or creatinine clearance > 60 mL/min
* Total serum bilirubin < 1.5 mg/dL
* Fertile patients must use effective contraception
* History of a curatively treated malignancy from which the patient has been disease-free for ≥ 2 years and has a survival prognosis of > 5 years

Exclusion Criteria:

* Pregnant or breast-feeding.
* Prior severe infusion reaction to a monoclonal antibody
* prior therapy specifically and directly targeting the epidermal growth factor receptor (EGFR) pathway
* Hypertension
* Uncontrolled diabetes
* Intercurrent illness that would likely interfere with protocol therapy or prevent surgical resection
* Any of the following within the past 6 months:

  * New York Heart Association class III-IV congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Unstable angina or myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10-02 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K. Gibson, MD, Study Chair — University of Pittsburgh
Locations (109):
- United States (109):
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - La Grange Oncology Associates - Geneva, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between June 10, 2008 and January 8, 2010. The first patient was accrued on October 2, 2008.
Period: Overall Study
Arm/Group | Neoadjuvant Therapy, Surgery, Adjuvant Therapy
Started | 22
Eligible and Began Treatment | 21
Underwent Surgery | 17
Received Adjuvant Therapy | 12
Completed | 9
Not Completed | 13
Not completed — Adverse Event | 7
Not completed — Death | 5
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Neoadjuvant Therapy, Surgery, Adjuvant Therapy
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 62 [45 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Pathologic Complete Response
Description: After neoadjuvant therapy, participants underwent surgical resection. The excised tumor was examined by a pathologist. A pathologic complete response is defined as the absence of any histopathologic evidence of tumor in the resected esophageal and nodal tissue specimen.
Time Frame: At time of surgery (which occurred 63 to 91 days after study entry)
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: Proportion of patients
Arm/Group | Neoadjuvant Therapy, Surgery, Adjuvant Therapy
Number analyzed (Participants) | 21
Proportion of patients | 0.33 [0.168 to 0.536]

ADVERSE EVENTS:
Time Frame: Assessed every 6 weeks while on treatment and for 30 days after the end of treatment
Groups:
- Neoadjuvant Therapy, Surgery, Adjuvant Therapy: 35 days of neoadjuvant chemoradiotherapy with oxaliplatin and infusional 5-fluorouracil plus cetuximab followed by post-operative docetaxel and cetuximab.
Arm/Group | Neoadjuvant Therapy, Surgery, Adjuvant Therapy
Serious Adverse Events (participants affected / at risk) | 19/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Therapy, Surgery, Adjuvant Therapy (N=22)
Allergic reaction (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 4
Leukocytes decreased (Investigations) | 2
Lymphopenia (Investigations) | 5
Neutrophils decreased (Investigations) | 1
Platelets decreased (Investigations) | 2
Heart block asystole (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac troponin I (cTnI) increased (Investigations) | 1
Hypotension (Vascular disorders) | 2
Fatigue (General disorders) | 5
Weight loss (Investigations) | 1
Activated partial thromboplastin time pr (Investigations) | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Coagulation-other (Investigations) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Radiation dermatitis (Injury, poisoning and procedural complications) | 1
Death - multiorgan failure (General disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 5
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 8
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4
Distention/bloating, abdominal (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 3
Esophagitis (Gastrointestinal disorders) | 5
Malabsorption (Gastrointestinal disorders) | 1
Muco/stomatitis (symptom) esophagus (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Necrosis, small bowel NOS (Gastrointestinal disorders) | 1
Perforation, colon (Gastrointestinal disorders) | 1
Stenosis (incl anastomotic) esophagus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Surgical hemorrhage (Injury, poisoning and procedural complications) | 1
Infection Gr0-2 neut, brain (Infections and infestations) | 1
Infection Gr0-2 neut, colon (Infections and infestations) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 1
Infection Gr0-2 neut, sm bowel (Infections and infestations) | 1
Infection w/ unk ANC wound (Infections and infestations) | 2
Infection Gr0-2 neut, blood (Infections and infestations) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Alkaline phosphatase increased (Investigations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Laryngeal nerve dysfunction (Nervous system disorders) | 1
Neuropathy-motor (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 1
Esophagus, pain (Gastrointestinal disorders) | 1
(ARDS) (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Therapy, Surgery, Adjuvant Therapy (N=22)
Anemia (Blood and lymphatic system disorders) | 16
Leukocytes decreased (Investigations) | 5
Lymphopenia (Investigations) | 3
Neutrophils decreased (Investigations) | 6
Platelets decreased (Investigations) | 9
Palpitations (Cardiac disorders) | 2
Hypotension (Vascular disorders) | 2
Fatigue (General disorders) | 18
Fever w/o neutropenia (General disorders) | 5
Insomnia (Psychiatric disorders) | 3
Weight loss (Investigations) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3
Nail changes (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 9
Radiation dermatitis (Injury, poisoning and procedural complications) | 5
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 10
Constipation (Gastrointestinal disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 11
Dysphagia (Gastrointestinal disorders) | 3
Esophagitis (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 4
Muco/stomatitis (symptom) esophagus (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 15
Salivary (Gastrointestinal disorders) | 3
Taste disturbance (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 11
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Edema limb (General disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Alkaline phosphatase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Acidosis (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 4
Dizziness (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 3
Neuropathy-motor (Nervous system disorders) | 3
Neuropathy-sensory (Nervous system disorders) | 11
Abdomen, pain (Gastrointestinal disorders) | 2
Chest/thoracic pain NOS (General disorders) | 2
Esophagus, pain (Gastrointestinal disorders) | 4
Head/headache (Nervous system disorders) | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 4
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No